CLINICAL TRIAL: NCT03342846
Title: The Effect of High Versus Low Frequency Repetitive Transcranial Magnetic Stimulation on Motor Dysfunction in Parkinson's Disease; Which is More Beneficial?
Brief Title: High Versus Low Frequency rTMS on Motor Dysfunction in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: High versus low TMS in PD.
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Frequency rTMS in PD (Active Comparator): The first group received 20 Hz rTMS on M1 daily for 10 days 5 sessions every week.
  Interventions: Device: rTMS
- Low Frequency rTMS in PD (Active Comparator): The second group received 1 Hz rTMS on M1 daily for 10 days 5 sessions every week.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — the first group received 20 Hz and the 2nd group received 1 Hz rTMS daily for 10 days 5 sessions every week on M1.

SUMMARY:
The aim of the study is to compare high versus low frequency rTMS on motor dysfunction in PD. Forty patients with PD participated in the study.

The patients were randomly assigned into two groups; the first group received 1Hz and the 2nd one received 20 Hz rTMS daily for 10 days 5 sessions every week. The doctors who assess the patients clinically is blind for the frequency of rTMS, also patients don't know which type of stimulation they received. The patients were followed up before and after the 10 sessions and one month later.

DETAILED DESCRIPTION:
The aim of the study is to compare high versus low frequency rTMS on motor dysfunction in PD. Forty patients with PD participated in the study.

The patients were randomly assigned into two groups; the first group received 1Hz and the 2nd one received 20 Hz rTMS daily for 10 days 5 sessions every week and 2 days off per week. The doctors who assess the patients clinically is blind for the frequency of rTMS, also patients don't know which type of stimulation they received. The patients were followed up before and after the 10 sessions and one month later.

ELIGIBILITY:
Inclusion Criteria:

* All PD patients who were diagnosed according to UK bank criteria for PD.

Exclusion Criteria:

* History of repeated head injury.
* History of repeated cerebrovascular strokes
* History of defined encephalitis
* Oculogyric crisis, supra nuclear gaze palsy.
* Family history of more than one relative
* severe dementia, MMSE < 23, severe depression
* Cerebellar signs
* Babiniski sign
* Hydrocephalus or intracranial lesion on neuroimaging
* Patients with intracranial on neuroimaging
* Patients with intracranial metallic device or pacemaker
* Patients who were unable to give informed consent because of severe anesthesia, or cognitive deficit

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
change in motor disability | one month
  Measure the change in motor disability by using UPDRS and self assessment scale

SECONDARY OUTCOMES:
Changes in Cortical excitability | Two weeks
  Measure the changes in cortical excitability using magnetic stimulation appratus

CONTACTS AND LOCATIONS:
Overall Officials: eman M Khedr, MD, Principal Investigator — Professor of Neurology, Faculty of Medicine, Assiut University
Locations (1):
- Eman Khedr, Asyut, Egypt